CLINICAL TRIAL: NCT03764345
Title: Sofosbovir/Ledipasvir in HCV Infected Children Aged From 4 to 10 Years
Brief Title: Eight Weeks Sofosbovir/Ledipasvir in HCV Infected Children Aged 4 to 10 Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Liver Institute, Egypt (Other)
Responsible Party: Principal Investigator, Mostafa M. Sira, Assistant Professor, National Liver Institute, Egypt
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sof-Led-HCV-Ped
Record Dates: First submitted 2018-11-28; First posted 2018-12-05 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Hepatitis C, Chronic; Children, Only
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sofosbovir/Ledipasvir Daily (Experimental): Patients receive oral daily dose of Sofosbovir/Ledipasvir (200/45mg) daily for 8 weeks
  Interventions: Drug: Sofosbovir/Lepipasvir (200/45mg) tablet (Heterosofir)

INTERVENTIONS:
Drug: Sofosbovir/Lepipasvir (200/45mg) tablet (Heterosofir) — Patients receive oral daily dose of Sofosbovir/Ledipasvir (200/45mg) daily for 8 weeks

SUMMARY:
Recently the era of direct-acting antiviral drugs for hepatitis C treatment has changed the world map of HCV. Results in adults are promising. FDA approved only two drugs in the pediatric age group 12 to 17 years. Younger children are still on the wait list for treatment. The current study aimed to treat children aged between 3 and 12 years with half the adult dose of Sofosbuvir/Ledipasvir combination (Heterosofir).

DETAILED DESCRIPTION:
The WHO has declared hepatitis C a global health problem, with ∼ 3% of the world's population (roughly 170-200 million individuals) infected with HCV. Egypt has the highest prevalence of HCV in the world, ranging from 6 to 28%, with an average of ∼ 13.8% in the general population. Ap-proximately 90% of Egyptian HCV isolates belong to a single subtype, 4a.

Hepatitis C virus (HCV) is a major cause of chronic liver disease and a prin-cipal reason for liver transplant; approximately 170 million people worldwide are chronically infected. There is general consensus that HCV elimination is associated with strong and sustained CD4+ and CD8+ T cell res-ponses that target multiple epitopes within the different HCV proteins, however, they are not maintained in patients who develop chronic disease . A variety of factors purportedly contribute to the dimi-nished T cell responses observed in chronically infected patients, including an im-paired dendritic cell (DC) function.

The successful development of direct-acting antivirals (DAAs) that are active against hepatitis C virus has transformed chronic hepatitis C infection from a con-dition requiring complex therapies with unsatisfactory outcomes to one that can be easily treated with few contraindications and side-effects. Since 2011, the US Food and Drug Administration (FDA) and the European Medicines Agency (EMA) have approved eight oral DAA regimens for the treatment of adults with chronic hepatitis C. Investigation into DAAs for children has been slower.

For adolescents aged 12-17 years, the safety and efficacy of the fixed-dose combination sofosbuvir and ledipasvir for genotype 1 or 4 infection and of combination sofosbuvir plus ribavirin for genotype 2 or 3 infection have been described in full-length articles.

A recent study explored the safety and efficacy of combination sofosbuvirplus ribavirin in Pakistani children (aged 5-18 years) with hepatitis C virus genotype 1, 2, or 3 infection. Further results have been presented as ab-stracts for the fixed-dose combination sofosbuvir and ledipasvir in children aged 6-11 years for the fixed-dose combination ombitasvir, pari-taprevir, and ritonavir with or without dasabuvir and with or without ribavirin in adolescents aged 12-17 years with genotype 1 or 4 infection and for combination sofosbuvir plus daclatasvir with or without ribavirin in Egyp-tian adolescents aged 12-17 years with genotype 4 infection.

Dendritic cells are professional antigen presenting cells characterized by a po-tent capacity to elicit primary T cell responses. Two major subsets of DC can be identified from human peripheral blood: plasmacytoid (p) DC and conventional or myeloid (m) DC. Each subset represents 0.3-0.5% of the normal human peripheral blood mononuclear cell (PBMC) population.

ELIGIBILITY:
Inclusion Criteria:

* Children with chronic HCV
* age 3- 12 y old
* weight 17- 35kg
* Basal HCV viremia less than 6.8 log IU/mL
* Treatment-naive
* No cirrhosis

Exclusion Criteria:

* Patients with dual HBV and HCV infection or associated with chronic hepatitis other than chronic HCV
* age below 3 years or above 12 years
* body weight less than 17 or more than 35 Kg
* HCV/HIV coinfection.
* Patients with HCV infection and HCC.
* Patients with HCV infection and underlying cardiac comorbidities
* Decompensated patients with HCV
* Hypoalbuminemia of < 3.5g/dL.
* International normalised ratio (INR) >2.
* Advanced fibrosis scoring by transient elastography (F 4 broScan)
* Any concomitant malignancy.
* Parents' refusal for participation of their children in the study.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2019-07-02 (Actual)

PRIMARY OUTCOMES:
Side effect 1 Number of patients with fatigue | 8 weeks
  Number of patients with fatigue
Side effect 2 Number of patients with Headache | 8 weeks
  Number of patients with Headache
Side effect 3 Number of patients with nausea | 8 weeks
  Number of patients with nausea
Side effect 4 Number of patients with diarrhea | 8 weeks
  Number of patients with diarrhea
Side effect 5 Number of patients with insomnia | 8 weeks
  Number of patients with insomnia
Side effect 6 Number of patients with weakness | 8 weeks
  Number of patients with weakness
Side effect 7 Number of patients with bradycardia | 8 weeks
  Number of patients with bradycardia
Side effect 8 Number of patients with cough | 8 weeks
  Number of patients with cough
Side effect 9 Number of patients with myalgia | 8 weeks
  Number of patients with myalgia
Side effect 10 Number of patients with dysapnea | 8 weeks
  Number of patients with dysapnea
Side effect 11 Number of patients with irritability | 8 weeks
  Number of patients with irritability
Side effect 12 Number of patients with dizziness | 8 weeks
  Number of patients with dizziness
Side effect 13 Number of patients with depression | 8 weeks
  Number of patients with depression
Side effect 14 Number of patients with skin rash | 8 weeks
  Number of patients with skin rash

SECONDARY OUTCOMES:
HCV-RNA PCR by the end of therapy | 8 weeks
  HCV-RNA PCR at week 8
HCV-RNA PCR after 20 weeks for SVR | 20 weeks
  HCV-RNA PCR at week 20

OTHER OUTCOMES:
Treatment safety-1 Alanine transaminase serum level | 8 weeks
  Alanine transaminase serum level
Treatment safety-2 Aspartate transaminase serum level | 8 weeks
  Aspartate transaminase serum level
Treatment safety-2 Degree of liver fibrosis | 8 weeks
  Liver Stiffness measurement before and after end of therapy
Treatment tolerability-1 Patient height | 20 weeks
  measurement of Height
Treatment tolerability-2 Body weight | 20 weeks
  measurement of weight

CONTACTS AND LOCATIONS:
Overall Officials: Behairy E Behairy, Prof, Principal Investigator — National Liver Institute, Menoufia University; Hanaa A El-Araby, Prof, Study Director — National Liver Institute, Menoufia University; Mohamed A El-Guindi, Prof, Study Director — National Liver Institute, Menoufia University; Hosam M Basiouny, MD, Study Chair — National Liver Institute, Menoufia University; Ola A Fouad, MD, Study Chair — National Liver Institute, Menoufia University; Ayman M Marey, Prof, Study Chair — Faculty of Medicine, Zagazig University; Bassam A Ayoub, MD, Study Chair — National Liver Institute, Menoufia University
Locations (1):
- Pediatric Hepatology, Gastroenterology and Nutrition Department, National Liver Institute, Menoufia University, Shebin El-Koom, Menofiya, Egypt

REFERENCES:
- [Background] Balistreri WF, Murray KF, Rosenthal P, Bansal S, Lin CH, Kersey K, Massetto B, Zhu Y, Kanwar B, German P, Svarovskaia E, Brainard DM, Wen J, Gonzalez-Peralta RP, Jonas MM, Schwarz K. The safety and effectiveness of ledipasvir-sofosbuvir in adolescents 12-17 years old with hepatitis C virus genotype 1 infection. Hepatology. 2017 Aug;66(2):371-378. doi: 10.1002/hep.28995. Epub 2017 Jun 19. PMID 27997679
- [Background] Deuffic-Burban S, Mohamed MK, Larouze B, Carrat F, Valleron AJ. Expected increase in hepatitis C-related mortality in Egypt due to pre-2000 infections. J Hepatol. 2006 Mar;44(3):455-61. doi: 10.1016/j.jhep.2005.08.008. Epub 2005 Sep 15. PMID 16310281
- [Background] El-Sayed M, Hassany M, Asem N. A pilot study for safety and efficacy of 12 weeks sofosbuvir plus daclatasvir with or without ribavirin in Egyptian adoles-cents with chronic hepatitis C virus Infection. Journal of Hepatology 2017,66:S178
- [Background] El-Serag HB. Hepatocellular carcinoma and hepatitis C in the United States. Hepatology. 2002 Nov;36(5 Suppl 1):S74-83. doi: 10.1053/jhep.2002.36807. PMID 12407579
- [Background] Gowans EJ, Jones KL, Bharadwaj M, Jackson DC. Prospects for dendritic cell vaccination in persistent infection with hepatitis C virus. J Clin Virol. 2004 Aug;30(4):283-90. doi: 10.1016/j.jcv.2004.03.006. PMID 15163415
- [Background] Hashmi MA, Cheema HA. Effectiveness and Safety of Sofosbuvir in Treatment-NaiveChildren with Hepatitis C Infection. J Coll Physicians Surg Pak. 2017 Jul;27(7):423-426. PMID 28818165
- [Background] Indolfi G, Serranti D, Resti M. Direct-acting antivirals for children and adolescents with chronic hepatitis C. Lancet Child Adolesc Health. 2018 Apr;2(4):298-304. doi: 10.1016/S2352-4642(18)30037-3. Epub 2018 Feb 24. PMID 30169301
- [Background] Kamal SM, Madwar MA, Peters T, Fawzy R, Rasenack J. Interferon therapy in patients with chronic hepatitis C and schistosomiasis. J Hepatol. 2000 Jan;32(1):172-4. doi: 10.1016/s0168-8278(00)80207-x. No abstract available. PMID 10673085
- [Background] Murray KF, Balistreri W, Bansal S, Whitworth S, Evans H, Gonzalez-Peralta R, et al. Ledipasvir/sofosbuvir±ribavirin for 12 or 24 weeks is safe and effective in children 6-11 years old with chronic hepatitis C infection. Journal of Hepatology 2017,66:S57-S58
- [Background] O'Doherty U, Peng M, Gezelter S, Swiggard WJ, Betjes M, Bhardwaj N, Steinman RM. Human blood contains two subsets of dendritic cells, one immunologically mature and the other immature. Immunology. 1994 Jul;82(3):487-93. PMID 7525461
- [Background] Takaki A, Wiese M, Maertens G, Depla E, Seifert U, Liebetrau A, Miller JL, Manns MP, Rehermann B. Cellular immune responses persist and humoral responses decrease two decades after recovery from a single-source outbreak of hepatitis C. Nat Med. 2000 May;6(5):578-82. doi: 10.1038/75063. PMID 10802716
- [Background] Thorne C, Indolfi G, Turkova A, Giaquinto C, Nastouli E. Treating hepatitis C virus in children: time for a new paradigm. J Virus Erad. 2015 Jul 1;1(3):203-5. doi: 10.1016/S2055-6640(20)30500-8. PMID 27482412
- [Background] Wirth S, Rosenthal P, Gonzalez-Peralta RP, Jonas MM, Balistreri WF, Lin CH, Hardikar W, Kersey K, Massetto B, Kanwar B, Brainard DM, Shao J, Svarovskaia E, Kirby B, Arnon R, Murray KF, Schwarz KB. Sofosbuvir and ribavirin in adolescents 12-17 years old with hepatitis C virus genotype 2 or 3 infection. Hepatology. 2017 Oct;66(4):1102-1110. doi: 10.1002/hep.29278. Epub 2017 Aug 26. PMID 28543053
- [Background] Schulze Zur Wiesch J, Ciuffreda D, Lewis-Ximenez L, Kasprowicz V, Nolan BE, Streeck H, Aneja J, Reyor LL, Allen TM, Lohse AW, McGovern B, Chung RT, Kwok WW, Kim AY, Lauer GM. Broadly directed virus-specific CD4+ T cell responses are primed during acute hepatitis C infection, but rapidly disappear from human blood with viral persistence. J Exp Med. 2012 Jan 16;209(1):61-75. doi: 10.1084/jem.20100388. Epub 2012 Jan 2. PMID 22213804